CLINICAL TRIAL: NCT03754257
Title: Effects of Electrical Stimulation for Preventing Loss of Muscle Mass in Patients With SIRS, Sepsis and Septic Shock - Randomized, Controlled and Double-blind Clinical Trial
Brief Title: Effects of Electrical Stimulation for Preventing Loss of Muscle Mass in Patients With SIRS, Sepsis and Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Wellington Yamaguti, Wellington Pereira dos Santos Yamaguti, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3.999.139
Record Dates: First submitted 2018-10-24; First posted 2018-11-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Septic Shock; SIRS
Keywords: sepsis; septic shock; electrical stimulation
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Electrical Stimulation (Experimental): Experimental Electrical Stimulation for 40 minutos + conventional physiotherapy, during seven days.
  Interventions: Procedure: Experimental Electrical Stimulation; Other: Conventional Physiotherapy
- Sham Electrical Stimulation (Sham Comparator): Sham Electrical Stimulation for 40 minutes + conventional physiotherapy, during seven days.
  Interventions: Procedure: Sham Electrical Stimulation; Other: Conventional Physiotherapy

INTERVENTIONS:
Procedure: Experimental Electrical Stimulation — Experimental Electrical Stimulation (100Hz) during 40 minutes
  Arms: Experimental Electrical Stimulation
Procedure: Sham Electrical Stimulation — Sham Electrical Stimulation (5Hz) during 40 minutes
  Arms: Sham Electrical Stimulation
Other: Conventional Physiotherapy — Active and passive exercises, and walking.

SUMMARY:
Background: Electrical stimulation has been used in critical patients as an adjunct strategy of early rehabilitation. In septic or septic shock patients there are reports of only two studies in the literature, with conflicting results.

Objective: To evaluate the effects of electrical stimulation in the prevention of muscle mass loss in patients admitted to the ICU with systemic inflammatory response syndrome (SIRS), sepsis or septic shock.

Methods: This is a randomized, controlled, double-blind clinical trial. Thirty-six patients with a diagnosis of SIRS, sepsis or septic shock (including patients with sepsis due to the new coronavirus - COVID-19) will be randomly assigned to experimental group and sham group. They will be evaluated in relation to muscle mass, peripheral muscle strength and functional status. They will also be submitted to the collection of inflammatory, metabolic, damage and muscular trophism markers.

Expected results: Electrical stimulation is expected to be able to prevent loss of muscle mass in patients admitted to the ICU with SIRS, sepsis or septic shock. In addition, it is expected to be able to preserve strength in this population without increasing the pro-inflammatory or metabolic response.

DETAILED DESCRIPTION:
This is a randomized, controlled, double-blind clinical trial. Thirty-six patients with a diagnosis of SIRS, sepsis or septic shock (including patients with sepsis due to the new coronavirus - COVID-19) will be randomly assigned to experimental group and sham group.They will be evaluated in relation to muscle mass, peripheral muscle strength and functional status. They will also be submitted to the collection of inflammatory, metabolic, damage and muscular trophism markers.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the ICU with a diagnosis of SIRS, sepsis or septic shock,
* aged ≥ 18 years,
* body mass index (BMI) ≤ 35 kg / m2,
* without diabetic polyneuropathy,
* without cardiac pacemaker,
* without diagnosis of neuromuscular diseases,
* absence of skin lesions.

Exclusion Criteria:

* heart attack,
* death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Muscle mass | 8 days
  Cross-sectional area
Muscle mass | 8 days
  Thickness

SECONDARY OUTCOMES:
Peripheral muscle strength | 8 days
  Medical Research Council Scale will be used to measure the peripheral muscle strength. The patient's effort is graded on a scale of 0-5:
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed. The total score ranges from 0 (complete tetraparesis) to 60 points (normal muscle strength).
Functional status | 8 days
  Functional status will be assessed using the Surgical Intensive Care Unit Optimal Mobilization Score. This score classifies mobility from 0 to 4:
  The SOMS "0 - No mobility" indicates that no mobilization should be considered due to the patients' clinical status.
  SOMS "1 - Passive mobilization" indicates that passive mobilization can be carried out in bed.
  SOMS "2 - Sitting" demonstrates that the patient is already able to sit on the bed or in a chair.
  SOMS "3 - Standing", indicates that the patient can perform orthostatism, with or without assistance.
  The highest level of SOMS "4 - Ambulation", shows that the patient is capable of ambulation.
Inflammatory | 5 days
  IL-1α
Inflammatory | 5 days
  IL-6
Inflammatory | 5 days
  IL-8
Inflammatory | 5 days
  IL-10
Inflammatory | 5 days
  IL-15
Inflammatory | 5 days
  MIP-1α
Inflammatory | 5 days
  TNF-α
Inflammatory | 5 days
  CRP
Metabolic, damage and muscular trophism markers | 5 days
  Lactate
Metabolic, damage and muscular trophism markers | 5 days
  CPK
Metabolic, damage and muscular trophism markers | 5 days
  IGF-1

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No